CLINICAL TRIAL: NCT00191594
Title: Open-Label Duloxetine Extension Phase in Patients Who Have Completed the HMDG Clinical Trial
Brief Title: Open-Label Duloxetine Extension Phase in Patients Who Have Completed Previous Duloxetine Trials
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9548; F1J-XM-HMED
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-01-26 (Estimated); Status verified 2007-01

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Duloxetine Hydrochloride

INTERVENTIONS:
Drug: Duloxetine Hydrochloride

SUMMARY:
A study in patients with depression

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients at least 18 years of age who have previously completed satisfactorily the Lilly sponsored previous clinical trial, and who are clinically controlled with Duloxetine, as judge by the investigator
* All females must test negative for a urine pregnancy test at Visit 1. Females of childbearing potential (not surgically sterilized and between menarche and 1 year postmenopausal) must agree to utilize medically acceptable and reliable means of birth control as determined by the investigator during the study. Women who are pregnant or breast-feeding may not participate in the study.
* Must sign the informed consent document (ICD).

Exclusion Criteria:

* Have received treatment within the last 30 days with a drug ( not including study drug) that has not received regulatory approval for any indication at the time of study entry.
* Patients who have entered the optional tapering period of the previous study.
* In the opinion of the investigator, patients judged to be at serious suicidal risk.
* Treatment with a MAOI within 14 days prior to Visit 1 or potential need to use MAOI during the study or within 5 days of discontinuation of the study drug.
* Any patient who previously experienced a serious adverse event while taking duloxetine unless approved by the Lilly Physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105
Dates: Start 2005-03; Study Completion 2006-08

PRIMARY OUTCOMES:
Adverse events

SECONDARY OUTCOMES:
Vital signs

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT- 5 hours, EST), Study Director — Eli Lilly and Company
Locations (6):
- Spain (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ourense
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salamanca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santiago de Composte
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zamora